CLINICAL TRIAL: NCT02275143
Title: Feasibility of Computed Tomography (CT) Coronary Angiogram Evaluation in Cancer Patients Having CT Thorax, Abdomen and Pelvis (CT TAP)
Brief Title: Computed Tomography (CT) Coronary Angiogram Evaluation in Cancer Patients Having CT Thorax, Abdomen and Pelvis
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/P/152
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Stenosis
Keywords: Computed Tomography of Thorax, Abdomen and Pelvis; cancer patients; coronary angiogram evaluation
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT TAP scan: Suitable patients will be identified after consultant radiologists have approved a request for cancer routine CT TAP scan.
  Interventions: Radiation: CT TAP Scan

INTERVENTIONS:
Radiation: CT TAP Scan — Modification of chest CT protocol in the routine CT TAP: The Research CT of Thorax will be acquired as per the routinely performed CTCA with inclusion of the lung apices. Therefore the study will be acquired axially with prospective gating.

SUMMARY:
Currently patients with certain cancer usually have routine follow up (Computed Tomography of Thorax, Abdomen and Pelvis) CT TAP scans to see response to treatment or relapse. The study proposal allows the evaluation of the coronary arteries by modifying the current CT TAP technique without significant additional procedures, intravenous contrast or radiation - i.e. an opportunistic Computed Tomography Coronary Angiogram (CTCA) without any penalty. The question is does performing Computed Tomography (CT) of the thorax in such a way confer important additional information about cardiac risk? At the same time the investigators need to ensure that doing scan as per CTCA protocol produces equivalent image quality to evaluate other structures in the chest. A recent small retrospective study has using a similar technique suggests that it may in fact improve image quality due to less cardiac related motion artefact.

DETAILED DESCRIPTION:
The study is a non-inferiority observational study to primarily ensure that the Computed Tomography of Thorax, Abdomen and Pelvis (CT TAP) technique produces equivalent image quality of the lungs (hence the need to scan with both conventional technique and the Electrocardiograph [ECG] gated technique) and secondarily to evaluate the effectiveness of demonstrating the coronary arteries in this cohort of patients who have not received heart rate control.

ELIGIBILITY:
Inclusion Criteria:

* Patients having routine follow up cancer CT TAP scan
* Age more than or equal to 40 years of age at the time of scan.
* Able to provide informed written consent
* Able to hold their breath for at least 10 seconds
* Has regular heart rate
* Able to follow verbal commands for breath holding and remain still for the duration of scanning
* Able to lie supine for the entirety of the scan

Exclusion Criteria:

* Patient unable to give informed consent.
* Patients unable to lie supine
* Patient not able to breath hold for at least 10 seconds.
* Patients not having regular heart rate. Patient with atrial fibrillation or >2 atrial or ventricular premature beats on a preoperative 12 lead ECG (suboptimal image quality results from irregular heart rhythms)
* Patient having eGFR <30, to avoid risk of contrast nephrotoxicity in patients potentially at risk) or chronic renal failure on dialysis
* Patient has known contrast reaction.
* Patient is pregnant.
* Patients BMI>35
* Unavailability of research slot to accommodate for the urgency of the scan requested.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having routine follow up cancer CT TAP scan
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Objective Image quality analysis | 20 minutes
  Calculating image noise as measured by standard deviation (SD) in a region of interest.
Objective Image quality analysis | 20 minutes
  Calculating contrast-to-noise ratio (CNR)
Subjective Image quality analysis | 20 minutes
  All image data sets will be presented in blinded and randomized manner to two experienced consultant radiologists. Subjective image quality will be assessed in terms of subjective image noise, subjective image contrast, lesion conspicuity, diagnostic confidence and artefacts. The image quality attributes are taken from the European Guidelines on Quality Criteria for Computerized Tomography document and have been proven to be robust in comparing subjective image quality.

SECONDARY OUTCOMES:
Dose estimation | 20 minutes
  The total exam dose-length product (DLP) displayed by the CT scanner at the end of each CTPA is recorded. The effective dose in mSv is calculated by multiplying the total DLP for each exam by the conversion coefficient for the chest of 0.014 (as taken from National Radiological Protection Board Document).
Coronary segments analysis | 20minutes
  Image quality of the 4 main coronary arteries (left main, left anterior descending, left circumflex, and right coronary artery) was determined based on a 4-point grading system - Non-diagnostic; Adequate; Good; Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Roobottom, MBChB FRCP, Study Director — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust (PHNT), Plymouth, Devon, United Kingdom